CLINICAL TRIAL: NCT04033029
Title: Antibiotic Plasma Concentrations During Continuous Renal Replacement Therapy With a High Adsorption Membrane (oXiris®)
Status: Completed | Type: Observational
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Helena Colom Codina, Principal Investigator, Hospital Universitari de Bellvitge
Other Study IDs: HCC-PIP-2018-01
Record Dates: First submitted 2019-02-20; First posted 2019-07-25 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Hemodiafiltration; Sepsis; Acute Kidney Injury
Keywords: Acute kidney Injury; Sepsis; Antibiotic plasma level; CRRT; oXiris®
MeSH Terms: conditions — Sepsis; Acute Kidney Injury | interventions — Continuous Renal Replacement Therapy; Anti-Bacterial Agents; Piperacillin, Tazobactam Drug Combination; Ceftazidime; Cefepime; Daptomycin; ceftolozane, tazobactam drug combination

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, ultrafiltrate and urine samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Patients under CVVHDF with high adsorption membrane: Continuous venovenous hemodiafiltration mode (CVVHDF) using PrismafleX eXeed™ system and high adsorbent polyethyleneimide membrane (oXiris®). Filtration parameters will be determined following the local protocol (dose of 25-30 ml/kg/h).
  Interventions: Device: Continuous venovenous hemodiafiltration with high adsorption membrane (oXiris®); Drug: Antibiotics

INTERVENTIONS:
Device: Continuous venovenous hemodiafiltration with high adsorption membrane (oXiris®) — CRRT initiation will be determined by the treating physician on charge, according with the current recommendations of clinical practice and prescriptions of CRRT and local management protocols. The CVVHDF mode will be performed by using PrismafleX eXeed™ system and high adsorbent polyethyleneimide membrane (oXiris®). Filtration parameters will be determined following the local protocol (dose of 25-30 ml/kg/h).
Drug: Antibiotics — Antibiotic concentration-time data will be collected and analyzed.
  Other Names: Piperacillin/tazobactam; Ceftazidime; Cefepime; Daptomycin; Ceftolozane/tazobactam

SUMMARY:
* Study: Open label, non-randomized, observational, descriptive and prospective pharmacokinetic.
* Patients: sepsis patients undergoing continuous renal replacement therapy (CRRT) and admitted at the Intensive care unit of Bellvitge University Hospitals. No power calculations needed.
* Antibiotic treatment: piperacillin, ceftazidime, cefepime, ceftolozane and daptomycin as their standard of care and doses will be at the discretion of the treating physician.
* CRRT treatment: continuous venovenous hemodiafiltration (CVVHDF) will be performed by using the PrismafleX eXeed™ system with a high adsorbent membrane (oXiris®).
* Antibiotic concentrations: blood pre and post filter, urine and ultrafiltrate samples will be collected at steady state conditions. Samplig time will depend on dosage regimens of each antibiotic.

DETAILED DESCRIPTION:
The study is an open label, non-randomized, observational, descriptive and prospective pharmacokinetic study.

Setting: this study will be conducted at the Intensive Care Unit at the Bellvitge University Hospital.

Study aims: the primary objective is to determine the PK/PD target attainment of piperacillin, ceftazidime, cefepime, ceftolozane and daptomycin in septic critically ill patients treated with CVVHDF using oXiris® membrane. Secondary aims are: i) to characterize the PK of piperacillin, ceftazidime, cefepime, ceftolozane and daptomycin in critically ill patients under CVVHDF therapy using oXiris® membrane by developing a population PK model; ii) to identify the clinical and demographic sources of PK variability observed in these patient and iii) to develop individualized dosing recommendations based on the PK/PD index associated with therapy success.

Recruitment process: patients who meet the inclusion criteria will be enrolled for at least 72 hours (maximum 96 hours).

Sample size: no power calculations are required for this study as it aims to investigate the PK of these antibiotics and does not intend to measure the effect of an intervention between two groups.

Antibiotic treatment: patients will receive piperacillin, ceftazidime, cefepime, ceftolozane/tazobactam or daptomycin as their standard of care. Doses will be at the discretion of the treating physician. At the same time, patients will be treated under continuous renal replacement techniques (CRRT) with continuous venovenous hemodiafiltration mode (CVVHDF) using PrismafleX eXeed™ system and high adsorbent polyethyleneimide membrane (oXiris®). Filtration parameters will be determined following the local protocol (dose of 25-30 ml/kg/h) CRRT initiation will be determined by the treating physician on charge, according with the current recommendations of clinical practice and prescriptions of CRRT and local management protocols. The decision to stop the treatment will be determined by:

* Adequate renal recovery status: adequate capacity to effectively maintain fluid and electrolyte homeostasis and urinary output (>450 ml in 24 h) without the use of diuretics.
* Hemodynamic stability without renal function recovery. Therapy will be continued as intermittent hemodialysis.

Antibiotic concentrations: blood, either pre and post filtration through oXiris® membrane, urine and ultrafiltrate samples will be obtained. Samples will be collected at 1) steady state conditions and 2) after minimum 24h from the concomitant administration of CRRT and antibiotic for piperacillin, ceftazidime, cefepime, ceftolozane and 48h for daptomycin. Sampling times will depend on the dosage regimen of each antibiotic therapy. Drug concentrations will be determined using a previously developed and validated measurement procedure based on ultra-high performance liquid chromatography-tandem mass spectrometry.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the setting of sepsis and requirements of CRRT with high adsorption membranes for at least 48 h
* Age >18 years
* Treatment with piperacillin, ceftazidime, cefepime, ceftolozane and daptomycin prescribed at the discretion of the treating intensive care physician.
* Written informed consent will be required before the inclusion of a patient whenever possible and will be requested from the nearest relatives in the other cases.

Exclusion Criteria: none.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients under continuous venovenous hemodiafiltration (CVVHDF) by using the PrismafleX eXeed™ system with a high adsorbent membrane (oXiris®) and requiring antibiotic treatment with: piperacillin, ceftazidime, cefepime, ceftolozane/tazobactam or daptomycin.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Number of individuals attaining a defined pharmacokinetic-pharmacodynamic target for antimicrobial therapy | 01/08/2019 - 31/12/2021
  Time above minimum inhibitory concentration (%fT > k× MIC) for betalactams, and total-drug AUC24/MIC ≥ 666 for daptomycin

SECONDARY OUTCOMES:
Antibiotic concentration-time data. | 01/08/2019 - 31/12/2021
  Antibiotic concentration-time data will be collected and analysed to characterize the PK profile of piperacillin, ceftazidime, cefepime, ceftolozane and daptomycin in critically ill patients under CRRT therapy using oXiris® membrane and a population PK model will be developed.
Blood flow (mL/min). CRRT covariate that can affect drug exposure and PK parameters. | 01/08/2019 - 31/12/2021
  Effect of CRRT settings, physiopathological and demographic data on drug exposure and PK parameters.
Dialysate flow rate (L/h). | 01/08/2019 - 31/12/2021
  CRRT covariate that can affect drug exposure and PK parameters. For each antibiotic, a population pharmacokinetic model will be developed.
Ultrafiltrate flow rate (L/h). | 01/08/2019 - 31/12/2021
  CRRT covariate that can affect drug exposure and PK parameters. For each antibiotic, a population pharmacokinetic model will be developed.
Replacement fluid (mL/h). | 01/08/2019 - 31/12/2021
  CRRT covariate that can affect drug exposure and PK parameters. For each antibiotic, a population pharmacokinetic model will be developed.
Extraction rate (L/h). | 01/08/2019 - 31/12/2021
  CRRT covariate that can affect drug exposure and PK parameters. For each antibiotic, a population pharmacokinetic model will be developed.
Urine output (mL/day). | 01/08/2019 - 31/12/2021
  Physiopathological variables that can affect drug exposure and PK parameters. For each antibiotic, a population pharmacokinetic model will be developed.
Albumin (g/L). | 01/08/2019 - 31/12/2021
  Physiopathological variables that can affect drug exposure and PK parameters. For each antibiotic, a population pharmacokinetic model will be developed.
Weight (Kg). | 01/08/2019 - 31/12/2021
  Physiopathological variables that can affect drug exposure and PK parameters. For each antibiotic, a population pharmacokinetic model will be developed.
Admission diagnosis: surgical, medical, trauma. | 01/08/2019 - 31/12/2021
  Physiopathological variables that can affect drug exposure and PK parameters. For each antibiotic, a population pharmacokinetic model will be developed.
Dosage (mg, frequency of administration and mode of administration) needed to achieve the PK/PD target. | 01/08/2019 - 31/12/2021
  Monte-Carlo Simulations using the population PK parameters of the final models in order to generate concentration-time profiles of n hypothetical subjects per dosing regimen will be performed. With this data, we will calculate the probability of target attainment of the PK/PD indices associated to antibiotic therapy success, which will translate in the development of individualized dosing recommendations for our patient population.

CONTACTS AND LOCATIONS:
Overall Officials: Helena Colom Codina, Phd, Principal Investigator — Universitat Autònoma de Barcelona
Locations (1):
- Helena Colom Codina, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vincent JL, Rello J, Marshall J, Silva E, Anzueto A, Martin CD, Moreno R, Lipman J, Gomersall C, Sakr Y, Reinhart K; EPIC II Group of Investigators. International study of the prevalence and outcomes of infection in intensive care units. JAMA. 2009 Dec 2;302(21):2323-9. doi: 10.1001/jama.2009.1754. PMID 19952319
- [Background] Brun-Buisson C. The epidemiology of the systemic inflammatory response. Intensive Care Med. 2000;26 Suppl 1(Suppl 1):S64-74. doi: 10.1007/s001340051121. PMID 10786961
- [Background] Kollef MH, Sherman G, Ward S, Fraser VJ. Inadequate antimicrobial treatment of infections: a risk factor for hospital mortality among critically ill patients. Chest. 1999 Feb;115(2):462-74. doi: 10.1378/chest.115.2.462. PMID 10027448
- [Background] Zaragoza R, Artero A, Camarena JJ, Sancho S, Gonzalez R, Nogueira JM. The influence of inadequate empirical antimicrobial treatment on patients with bloodstream infections in an intensive care unit. Clin Microbiol Infect. 2003 May;9(5):412-8. doi: 10.1046/j.1469-0691.2003.00656.x. PMID 12848754
- [Background] Pinder M, Bellomo R, Lipman J. Pharmacological principles of antibiotic prescription in the critically ill. Anaesth Intensive Care. 2002 Apr;30(2):134-44. doi: 10.1177/0310057X0203000203. PMID 12002919
- [Background] Ibrahim EH, Sherman G, Ward S, Fraser VJ, Kollef MH. The influence of inadequate antimicrobial treatment of bloodstream infections on patient outcomes in the ICU setting. Chest. 2000 Jul;118(1):146-55. doi: 10.1378/chest.118.1.146. PMID 10893372
- [Background] Craig WA. Pharmacokinetic/pharmacodynamic parameters: rationale for antibacterial dosing of mice and men. Clin Infect Dis. 1998 Jan;26(1):1-10; quiz 11-2. doi: 10.1086/516284. PMID 9455502
- [Background] Roberts JA, Roberts MS, Robertson TA, Dalley AJ, Lipman J. Piperacillin penetration into tissue of critically ill patients with sepsis--bolus versus continuous administration? Crit Care Med. 2009 Mar;37(3):926-33. doi: 10.1097/CCM.0b013e3181968e44. PMID 19237898
- [Background] Heinemeyer G, Link J, Weber W, Meschede V, Roots I. Clearance of ceftriaxone in critical care patients with acute renal failure. Intensive Care Med. 1990;16(7):448-53. doi: 10.1007/BF01711224. PMID 2269714
- [Background] Trotman RL, Williamson JC, Shoemaker DM, Salzer WL. Antibiotic dosing in critically ill adult patients receiving continuous renal replacement therapy. Clin Infect Dis. 2005 Oct 15;41(8):1159-66. doi: 10.1086/444500. Epub 2005 Sep 12. PMID 16163635
- [Background] Carcelero San Martin E, Soy Muner D. [Dosage of antipseudomonal antibiotics in patients with acute kidney injury subjected to continuous renal replacement therapies]. Med Intensiva. 2013 Apr;37(3):185-200. doi: 10.1016/j.medin.2012.02.012. Epub 2012 Apr 3. Spanish. PMID 22475763
- [Background] Matzke GR, Frye RF, Joy MS, Palevsky PM. Determinants of ceftazidime clearance by continuous venovenous hemofiltration and continuous venovenous hemodialysis. Antimicrob Agents Chemother. 2000 Jun;44(6):1639-44. doi: 10.1128/AAC.44.6.1639-1644.2000. PMID 10817721
- [Background] Bauer SR, Salem C, Connor MJ Jr, Groszek J, Taylor ME, Wei P, Tolwani AJ, Fissell WH. Pharmacokinetics and pharmacodynamics of piperacillin-tazobactam in 42 patients treated with concomitant CRRT. Clin J Am Soc Nephrol. 2012 Mar;7(3):452-7. doi: 10.2215/CJN.10741011. Epub 2012 Jan 26. PMID 22282479
- [Background] Valtonen M, Tiula E, Backman JT, Neuvonen PJ. Elimination of meropenem during continuous veno-venous haemofiltration and haemodiafiltration in patients with acute renal failure. J Antimicrob Chemother. 2000 May;45(5):701-4. doi: 10.1093/jac/45.5.701. PMID 10797097
- [Background] Roberts DM, Roberts JA, Roberts MS, Liu X, Nair P, Cole L, Lipman J, Bellomo R; RENAL Replacement Therapy Study Investigators. Variability of antibiotic concentrations in critically ill patients receiving continuous renal replacement therapy: a multicentre pharmacokinetic study. Crit Care Med. 2012 May;40(5):1523-8. doi: 10.1097/CCM.0b013e318241e553. PMID 22511133
- [Result] Seyler L, Cotton F, Taccone FS, De Backer D, Macours P, Vincent JL, Jacobs F. Recommended beta-lactam regimens are inadequate in septic patients treated with continuous renal replacement therapy. Crit Care. 2011;15(3):R137. doi: 10.1186/cc10257. Epub 2011 Jun 6. PMID 21649882
- [Result] Rigo-Bonnin R, Ribera A, Arbiol-Roca A, Cobo-Sacristan S, Padulles A, Murillo O, Shaw E, Granada R, Perez-Fernandez XL, Tubau F, Alia P. Development and validation of a measurement procedure based on ultra-high performance liquid chromatography-tandem mass spectrometry for simultaneous measurement of beta-lactam antibiotic concentration in human plasma. Clin Chim Acta. 2017 May;468:215-224. doi: 10.1016/j.cca.2017.03.009. Epub 2017 Mar 10. PMID 28288784